CLINICAL TRIAL: NCT03312712
Title: Validation of the Analysis Methodology Behind the Use of Quantitative 2-deoxy-2-[Fluorine-18] Fluoro-D-glucose (18F-FDG) Positron Emission Tomography/Computed Tomography (PET/CT) to Assess Lung Inflammation
Brief Title: Validation of the Analysis Methodology Behind the Use of Quantitative 18F-FDG PET/CT to Assess Lung Inflammation
Acronym: VERIFY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Joseph Cheriyan, MD, Consultant Clinical Pharmacologist & Physician/Associate Lecturer, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: VERIFY
Record Dates: First submitted 2017-10-09; First posted 2017-10-18 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Lung Inflammation; Sarcoidosis
Keywords: FDG; PET; CT; Sarcoidosis
MeSH Terms: conditions — Pneumonia; Sarcoidosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples and Bronchoalveolar lavage (fluid taken as part of sarcoidosis patient standard of care bronchoscopy at Papworth Hospital) will be analysed at either Cambridge University Hospitals or Papworth Hospital.
  Research specific venous blood and urine samples will be also obtained, where applicable, as per the study protocol for all participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with sarcoidosis: * Bronchoscopy, BAL collection, and PFTs* [SoC] *if required
  * Screening, research and safety bloods
  * Dynamic 18F-FDG PET/CT scan
  Interventions: Radiation: PET/CT scan; Diagnostic Test: Blood and urine sampling
- Healthy volunteers: Part A:
  * PFTs
  * Screening, research and safety bloods
  * Dynamic 18F-FDG PET/CT scan
  Part B:
  * PFTs
  * Screening, research and safety bloods
  * Baseline and post challenge Dynamic 18F-FDG PET/CT scans
  * LPS/saline challenge
  Interventions: Radiation: PET/CT scan; Other: LPS Challenge; Other: Saline Challenge; Diagnostic Test: Blood and urine sampling

INTERVENTIONS:
Radiation: PET/CT scan — PET/CT will be performed at Cambridge University Hospital's PET-CT unit, Cambridge.
  Participants in Part A of the study (sarcoidosis and HVs) will receive one PET/CT scan. A Cine-CT scan will be performed immediately prior to the 18F-FDG PET/CT scan. Settings for the CT scans will be determined by clinical protocols, radiation dose will be kept as low as reasonably practicable (ALARP) consistent with UK legislation.
  After 6 hours of fasting and if blood glucose concentration is ≤11mmol/L participants will proceed to undergo an 18FDG PET/CT scan.
  18F-FDG will be administered intravenously at a dose of approximately 200 MBq.
  Positron emission scanning will involve a 60-minute dynamic acquisition from the lungs.
Other: LPS Challenge — In Part B, eight healthy volunteers will undergo an LPS challenge whereby each participant is injected with the challenge agent, Lipopolysaccharide (LPS), to invoke temporary mild lung inflammation. Each participant will have a PET/CT scan before and after the administration of LPS and the images will be assessed to determine whether these methods are able to detect true lung inflammation.
  Groups: Healthy volunteers
Other: Saline Challenge — In Part B, four healthy volunteers will undergo a saline challenge as outlined above for the LPS challenge. Pre- and post-challenge scans will provide control data for the study.
  Groups: Healthy volunteers
Diagnostic Test: Blood and urine sampling — For women whose post-menopausal status and/or pregnancy status is uncertain at screening, a blood sample will be collected to test for pregnancy and menopausal status (hormone profiling) before enrolling them on to the study. If pregnancy status is still uncertain at study visits, participants will have a urine pregnancy test before undergoing any PET/CT scans to ensure it is safe for them to continue in the study.

SUMMARY:
The purpose of this study is to validate the method of analysing Positron Emission Tomography (PET) images to assess lung inflammation. Development of novel therapeutic drugs requires a biomarker which is sensitive to the underlying disease and can respond to therapeutic interventions. PET is a potential imaging biomarker which can target molecular and cellular processes. There is currently no standardised method of analysing PET lung data and a lack of validation for the existing techniques.

This study is divided in to two parts. Part A aims to determine the best method to perform 18F-FDG PET/CT lung analysis and how it correlates with cell counts from bronchoalveolar lavage (BAL) samples taken from participants with active pulmonary sarcoidosis.

Part B will compare imaging data from healthy volunteers who have either undergone a Lipopolysaccharide (LPS) challenge (whereby the lung is temporarily inflamed) or saline equivalent to determine whether lung inflammation can be detected by 18F-FDG PET/CT. No medications will be given and patients will not be asked to stop or change existing medication.

DETAILED DESCRIPTION:
Inflammation plays an important role in a myriad of human diseases. Interstitial Lung Diseases (ILDs) are characterised by widespread inflammation and represent a major burden to the health sector. Imaging offers a method of assessing lung inflammation which is non-invasive and may help facilitate the development of new therapeutic drugs. Positron Emission Tomography (PET) is a sensitive imaging modality that uses radioactive material to highlight areas of disease. 18F-FDG is the most common radioactive tracer; it accumulates in cells with an increased metabolic rate. Previous studies have shown that inflammatory cells have an increased metabolic rate, thus PET imaging could highlight inflammation. 18F-FDG PET has been used in many studies exploring lung diseases; the concentration of tracer is thought to relate to the severity of inflammation.

There is currently no standardised method to analyse FDG-PET scans to assess the concentration of tracer in the lung (and therefore inflammation). A major challenge is providing corrections to ensure that the image only represents tracer in the lung tissue. Such corrections are non-trivial and affect how images are interpreted. A robust validation is needed to ensure that the analysis methods used in FDG-PET images truly represent the degree of lung inflammation.

Part A of this study aims to validate and compare the different analysis methods. Pulmonary sarcoidosis is a disease characterised by widespread lung inflammation. In Part A of the study the investigators will recruit patients with this condition, as well as age and gender matched (wherever possible) healthy volunteers. All Part A participants will receive one dynamic 18F-FDG PET/CT scan. The investigators will assess the uptake of 18FDG from PET images from patients with sarcoidosis versus those taken from healthy volunteers to validate and assess the reliability of the analysis method.

For Part B of the study the investigators will recruit healthy volunteers aged 50 or more. If sarcoidosis patients in Part A are 50 years old or more, the age-matched HV will be recruited in to Part B instead, thus potentially minimising the number of HVs that might need to be recruited in to Part A of the study.

The aims of this research study are:

i) To compare FDG-PET derived tissue inflammation measures against measures of inflammation from BAL samples.

ii) To compare different models of 18F-FDG lung analysis in patients with pulmonary sarcoidosis.

iii) To identify whether FDG PET is sensitive enough to detect a change in inflammation induced in healthy volunteers.

ELIGIBILITY:
For patients with sarcoidosis:

Inclusion Criteria:

* Suspected pulmonary sarcoidosis (as determined by referring physician)
* Requires bronchoscopy, EBUS and BAL (as determined by ILD team at Royal Papworth or Addenbrooke's Hospitals).
* Male or female ≥ 30 years with a BMI of 17-35kg/m2
* Consents to additional bronchoscopic evaluation during NHS mandated bronchoscopy, EBUS and BAL.

Exclusion Criteria:

* Inability to provide Informed Consent.
* A cardiovascular event in the last 6 months (i.e. acute coronary syndrome, unstable angina, CABG, PCI, stroke, MI, carotid endarterectomy).
* Patients with known clinically significant pulmonary diagnoses of COPD, lung fibrosis, interstitial lung disease, or α1-antitrypsin deficiency.
* Active smoking during the last 5 years.
* Patients with known chronic infections such as HIV or known active tuberculosis.
* Patients with rheumatoid arthritis, connective tissue disorders and other conditions known to be associated with active chronic inflammation (e.g. Inflammatory Bowel Disease).
* Known diabetes mellitus or known impaired glucose tolerance
* Participation in a previous research trial in the last three years which involved exposure to significant ionising radiation (i.e. cumulative research radiation dose >10 mSv)
* Pregnancy
* Women of childbearing potential [i.e. either postmenopausal or documented hysterectomy and/or bilateral oophorectomy - tubal ligation is not sufficient].
* Use of systemic steroids (oral or intravenous) at a dose > 10mg od of prednisolone or equivalent and/or antibiotics 4 weeks prior to PET/CT scan
* Any medical history or clinically relevant abnormality that is deemed by the principal investigator and/or medical monitor to make the subject ineligible for inclusion because of a safety concern

For healthy volunteers:

Inclusion criteria:

* Age/gender-matched group (Part A only): Male or female ≥ 30 years with a BMI of 17-35kg/m2 inclusive
* LPS/saline challenge group (Part B only): Male or female ≥ 50 years with a BMI of 17-35kg/m2 inclusive
* No smoking history
* Normal predicted spirometry values: FEV1/FVC > 0.7 and FEV1 > 80% predicted
* Healthy as determined by clinical history & examination by the investigator

Exclusion criteria:

* Inability to provide informed consent
* Pregnancy
* Patients with known chronic inflammation conditions such as rheumatoid arthritis, connective tissue disorders and inflammatory bowel disease
* A significant cardiovascular event in the last 6 months
* Insulin dependent diabetes mellitus or known impaired glucose tolerance
* Participation in previous research trial in the last three years which involves exposure to significant ionising radiation (cumulative dose >10mSv)
* Use of systemic steroids (oral or intravenous) at a dose > 10mg od of prednisolone or equivalent and/or antibiotics 4 weeks prior to PET/CT scan
* Any medical history or clinically relevant abnormality that is deemed by the principal investigator and/or medical monitor to make the subject ineligible for inclusion because of a safety concern
* Women of childbearing potential
* Patients with known chronic infections such as HIV or known active tuberculosis.
* Active smoking history (defined as > than 1 cigarette per day on a regular basis) over lifetime
* Known lung and/or respiratory disease or associated symptoms (e.g. dyspnoea, wheeze)

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort 1: Participants with suspected pulmonary sarcoidosis Cohort 2: Healthy volunteers who are non-smokers, age and gender matched, where possible, to cohort 1 participants
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2018-01-23 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Validation of 18F-FDG methodology used to assess lung inflammation in participants with sarcoidosis | Up to 4 weeks
  18F-FDG will be assessed using Patlak analysis and a compartmental model. This will be validated against histological samples from lung biopsies taken as part of the patient's standard clinical care prior to enrolling on to this study, and the inflammatory cell counts and densities (principally of macrophages and neutrophils) from BAL fluid in sarcoidosis patients.

SECONDARY OUTCOMES:
Pulmonary function tests | Screening Visit (V1)
  Spirometry (FVC and FEV1)
Pulmonary function tests | Screening Visit (V1)
  Gas transfer (TLCO measurement). Healthy volunteers will be asked to blow hard and fast into a mouthpiece for as long as possible and hold their breath for about 10 seconds.
Plasma biomarkers of inflammation | Up to 4 weeks
  CRP levels (mg/L)
Plasma biomarkers of inflammation | Up to 4 weeks
  Fibrinogen levels (mg/dL)
Leukocyte count and activity from BAL fluid samples | Up to 6 weeks
  Immunohistochemical staining where necessary (cell count)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cheriyan, MBChB, MA, FRCP, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Royal Papworth Hospital NHS Foundation Trust, Papworth Everard

IPD SHARING:
Plan to Share IPD: No